CLINICAL TRIAL: NCT04844398
Title: Effects of Clown Visits by RED NOSES Clowndoctors Austria on Stress and Mood in Children and Adolescents in Psychiatric Care - A Pilot Study
Brief Title: Clown Visits in Child and Adolescent Psychiatry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vienna (Other)
Collaborators: RED NOSES Clowndoctors Austria (Unknown)
Responsible Party: Principal Investigator, Martina Zemp, Prof. Dr., University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00675
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Subjective Stress; Mood States; Physiological Stress
Keywords: Pilot Projects; Art Therapy; Healthcare clowning; Humour; Child; Adolescent; Psychiatric care; Outpatients; Inpatients; Stress, Psychological; Saliva; Arousal; Mental Health Services; Delivery of Health Care
MeSH Terms: conditions — Subjective Stress; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Using a non-controlled pre-/post-test design, the level of salivary cortisol and self-reported stress and mood will be measured before and after each clown visit on a weekly basis over four consecutive weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clown visits (four times) (Experimental): Children and adolescents in psychiatric care participate in clown visits in a group setting on a weekly basis over four consecutive weeks.
  Interventions: Other: Clown visits by RED NOSES Clowndoctors Austria

INTERVENTIONS:
Other: Clown visits by RED NOSES Clowndoctors Austria — Participants will receive one clown visit per week over four weeks in a group setting. The visits will take place in at least two different wards of each participating psychiatric care facility. In each ward, max. 10 participants will be targeted. The visits are carried out routinely by two professional clown artists from RED NOSES Clowndoctors Austria. The duration of the visits and the specific artistic sequences will take place according to internally organized routines. The essence of the clown visit is to catch the patient's attention proactively and reach the highest level of engagement possible. The specific artistic sequences are implemented spontaneously according to the situational atmosphere and current mood of participants. One clown visit will last between 1 and 2 hours depending on age and number of participants. Each participant will be engaged between 5 and 10 minutes by the clown. The clown artists are not involved in any study-related research activities.

SUMMARY:
This pilot study aims at investigating short-term effects of clown visits by RED NOSES Clowndoctors Austria in children and adolescents in psychiatric care without control group. It is assumed that children and adolescents involved in an interaction with the clowns will experience a shift in their focus. Individual attention and distraction from painful emotions have the ability to redirect their attention to the current pleasurable moment and increase their level of energy. Scientific evidence has shown that the distraction and switch to positive emotions associated with healthcare clowning can decrease the level of stress and pain (Vagnoli et al., 2005; Dionigi et al., 2014).

The study examines subjective and physiological stress levels of participants receiving clown visits in a group setting on a weekly basis. Using a non-controlled pre-/post-test design, the level of salivary cortisol and self-reported stress and mood will be measured before and after each clown visit over four consecutive weeks. Additionally, effects on care staff at the health facilities will be assessed based on a questionnaire after each clown visit within the same time period of four weeks. The sample will consist of approximately 40 children and adolescents in inpatient or outpatient psychiatric care. The examined intervention, i.e. clown visits by RED NOSES Clowndoctors Austria, is an integral part within the selected psychiatric health care institutions.

The study hypotheses are:

1. Children and adolescents will report a reduced subjective stress level and better mood states in the three assessed dimensions (good - bad mood; alertness - tiredness; calmness - restlessness) after the experience of a clown visit (post-test) compared to before the clown visit (pre-test) independent of age and gender.
2. Children and adolescents will display a reduced cortisol level after the experience of a clown visit (post-test) compared to before the clown visit (pre-test) independent of age and gender.
3. The more frequently children and adolescents experience the weekly clown visits over the course of the four-week study, the stronger the stress-reducing and mood-enhancing effects in the pre-/post-comparison will be over time.
4. Self-reported perceptions of care staff at the health facilities will indicate a positive effect of the clown visits on their own individual moods, the atmosphere within the care team, and the patients' well-being.

DETAILED DESCRIPTION:
This pilot study will examine the effects of clown visits by RED NOSES Clowndoctors Austria on physiological and psychological stress indicators in approximately 40 children and adolescents aged between 7 and 18 years in Austrian inpatient or outpatient psychiatric health care institutions (without control group).

The data collection process will start with a baseline assessment on participants' general mental and physical health status, perceived stress, and coping with stress using standardized questionnaires. Subsequently, both salivary cortisol as well as self-reported stress and mood states of children and adolescents will be collected before and after each clown visit on a weekly basis over four consecutive weeks (pre-/post-test design). Saliva samples of cortisol are collected as a marker for the physiological stress response of participants. We will use Salicaps collection devices consisting of collection tubes and straws. Participants will be thoroughly instructed to collect accumulated saliva for two minutes without swallowing. After the two minutes, participants will transfer the accumulated saliva into the Salicap tube via the straw. Furthermore, self-reported stress levels and different dimensions of current mood states (good - bad mood; alertness - tiredness; calmness - restlessness) of children and adolescents are assessed by self-developed visual analogue scales and standardized questionnaires. In addition, representatives of the care staff at the health facilities will be asked to complete a questionnaire about their personal perception on the effects of clown visits on their own individual mood, the atmosphere within the care team, and the patients' well-being after each clown visit within the same time period of four weeks. The application of questionnaires is paper-based (paper-pencil). All data collected will be treated in a pseudonymized form.

Participants will be recruited from selected psychiatric health care facilities in Austria. The recruitment process of children and adolescents will be initiated by a briefing interview with the care staff at the relevant facilities. In this briefing, the staff will be informed in detail about the study goals and all data collection procedures and will have the opportunity to evaluate the participation of the children and adolescents independently (cf. eligibility criteria). No sensitive data will be shared with the research team at that point. The staff will further support in obtaining the written consent from parents or legal guardians prior to the start of data collection.

ELIGIBILITY:
Inclusion criteria:

1. Being aged between 7 and 18 years;
2. Currently being in inpatient or outpatient psychiatric treatment;
3. Regularly participating in clown visits at the relevant health facility;
4. A written consent of the child's legal guardian.

Exclusion criteria:

1. Potential negative impacts of clown visits or study participation on participants' health or well-being according to medical or paramedical care staff of the relevant health facility;
2. Insufficient command of German (for self-reports only).

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Subjective Stress | Pre-Post-Change: Change from before to immediately after intervention for four times (over four weeks)
  Subjective stress levels of children and adolescents will be assessed before as well as after each of the four clown visits by self-developed visual analogue scales (0-100 with higher scores indicating greater subjective stress).
Subjective Mood | Pre-Post-Change: Change from before to immediately after intervention for four times (over four weeks)
  Subjective mood states (good - bad mood; alertness - tiredness; calmness - restlessness) of children and adolescents will be assessed before as well as after each of the four clown visits by an adapted and shorted version of the "Multidimensional Mood Questionnaire" (Steyer et al., 1997).
Physiological Stress: Salivary Cortisol | Pre-Post-Change: Change from before to immediately after intervention for four times (over four weeks)
  Saliva samples of cortisol are collected as a marker for the physiological stress response of children and adolescents. Salivary cortisol reflects the activity of the HPA axis. Samples will be collected before as well as after each of the four clown visits. We will use Salicaps collection devices consisting of collection tubes and straws. Participants will be thoroughly instructed to collect accumulated saliva for two minutes without swallowing. After the two minutes, participants will transfer the accumulated saliva into the Salicap tube via the straw. Tubes are then stored at -20°C prior to analysis in the biochemical laboratory.
Evaluation of Care Staff | Post-assessment: after each of the four interventions
  Self-reported perceptions of care staff in the health facility will be assessed using a self-developed questionnaire about the effects of the clown visits on their own individual moods, the atmosphere within the care team, and the patients' well-being after each of the four clown visits.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline (before intervention)
  Children's and adolescents' self-reported health-related quality of life will be assessed at baseline by the revised questionnaire "Health-Related Quality of Life" (German version; Ravens-Sieberer & Bullinger, 1998).
Internalizing and Externalizing Symptoms | Baseline (before intervention)
  Children's and adolescents' self-reported emotional and behavioral problems will be assessed at baseline by the relevant subscales of the questionnaire "Strengths and Difficulties Questionnaire" (German version; Klasen et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Zemp Martina, PhD, Principal Investigator — University of Vienna; Simone Seebacher, Mag., Study Chair — RED NOSES Clowndoctors Austria; Maggie Rössler, PhD, Study Chair — RED NOSES Clowndoctors Austria; Urs Nater, PhD, Study Director — University of Vienna

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and syntaxes of this study will be made openly available in OSF Storage at https://osf.io/.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol including the SAP will become available before the start of data collection.
URL: http://osf.io/

REFERENCES:
- [Derived] Zemp M, Friedrich AS, Holzmeier L, Seebacher S, Rossler M, Nater UM. Effects of clown visits on stress and mood in children and adolescents in psychiatric care-Protocol for a pilot study. PLoS One. 2022 Feb 18;17(2):e0264012. doi: 10.1371/journal.pone.0264012. eCollection 2022. PMID 35180260